CLINICAL TRIAL: NCT03248583
Title: Decision-Making Processes While Online Grocery Shopping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Albany (Other)
Responsible Party: Principal Investigator, Julia Hormes, Assistant Professor of Psychology, University at Albany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-E-005-01
Record Dates: First submitted 2017-07-28; First posted 2017-08-14 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Nutrition Poor
Keywords: Proof-of-principle; Feasibility
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Default (Experimental)
  Interventions: Other: Default option
- Psychoeducation (Active Comparator)
  Interventions: Other: Psychoeducation
- Incentive (Active Comparator)
  Interventions: Other: Incentive

INTERVENTIONS:
Other: Default option — The "default option" is a behavioral economics construct that refers to the option a consumer selects if no active choice is made (e.g. opt-out 401K plans, which significantly increase enrollment, compared to active sign up).
  Participants in the default condition were presented with a pre-filled online shopping cart containing a combination of groceries that meet macro- and micronutrient requirements for their gender and age, and told that they are free to delete, add, and exchange any item they wish to finalize their selections.
  Arms: Default
Other: Psychoeducation — Participants in the psychoeducation condition were instructed to read a brief psychoeducational brochure adapted from materials currently utilized by the New York State Office of Temporary and Disability Assistance ("Eat Smart New York").
  Arms: Psychoeducation
Other: Incentive — Participants in the incentive condition were informed that they will receive a gift card to a major retailer of their choice if they select groceries that meet recommended nutritional guidelines for macro- and micronutrient requirements. Participants were given examples of macro- and micronutrients to ensure that the instructions were clear.
  Arms: Incentive

SUMMARY:
Individuals living with food insecurity are disproportionately affected by overweight and obesity and associated chronic health problems. There remains a lack of sustainable and scalable interventions targeting widespread barriers to access to healthy foods in this population to increase the nutritional quality of foods purchased for preparation and consumption at home.

This randomized controlled proof-of-principle trial was designed to examine the feasibility and initial efficacy of a "default option" in enhancing the nutritional quality of groceries selected via the online shopping service of a local grocery store under conditions that mimic the financial constraints typical of individuals living with food insecurity.

In behavioral economics, the "default option" refers to the option a consumer selects if no active choice is made. The notion of the default option is based on the concept of "asymmetrical" or "libertarian paternalism," which seeks to subtly shift consumer behavior in a manner that promotes welfare, but without overtly interfering with the individual's freedom to choose.

It was hypothesized that the "default" option effectively increases the nutritional quality of foods purchased online, compared to monetary incentives and psychoeducation about nutrition.

Female undergraduate students (n = 60) selected food for one week using the online shopping service of a local grocery store with a budget corresponding to maximum weekly Supplemental Nutrition Assistance Program (SNAP) benefits. Before completing the task again, participants were randomized to: (1) a small monetary "incentive" for selecting groceries that meet nutritional guidelines (n = 17), (2) an "educational" brochure (n = 24), or (3) a "default" pre-filled online shopping cart containing a nutritionally balanced selection of groceries to which they could freely make changes (n = 18).

Primary outcome measures capture the nutritional quality of groceries selected/ purchased.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* fluent in written and spoken English
* able to provide informed consent

Exclusion Criteria:

* significant dietary restrictions (i.e., meat avoidance, food allergies, religious dietary restrictions, etc.)
* likely presence of current eating disorder diagnosis (score >/= 2 on SCOFF screening measure)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility was based in part on self-representation of gender identity as female.
Enrollment: 60 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2016-09-29 (Actual); Study Completion 2016-09-29 (Actual)

PRIMARY OUTCOMES:
Nutritional quality | Single laboratory visit, <1.5 hours
  The Thrifty Food Plan Calculator (TFPC) was used to quantify the nutritional quality of groceries selected by study participants. The TFPC was developed using U.S. Department of Agriculture nutrition and consumption data and is designed to have users input information about the relative amount of money spent on various categories of food and provides comprehensive information on caloric, macro-, and micronutrient content of the foods selected based on participant age and gender.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Coffino JA, Hormes JM. A Default Option to Enhance Nutrition Within Financial Constraints: A Randomized, Controlled Proof-of-Principle Trial. Obesity (Silver Spring). 2018 Jun;26(6):961-967. doi: 10.1002/oby.22151. Epub 2018 Mar 31. PMID 29604181